CLINICAL TRIAL: NCT03676946
Title: An Open-label, Dose-escalation, Bi-weekly Phase I+II Clinical Trial in Treating Patients With Locally Advanced and Metastatic Urothelial Carcinoma
Brief Title: A Clinical Study of PD-L1 Antibody ZKAB001（Drug Code） in Locally Advanced and Metastatic Urothelial Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NTL-LEES-2017-01
Record Dates: First submitted 2018-09-13; First posted 2018-09-19 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZKAB001 5mg/kg (Experimental): Three or six patients will be treated with the dose of 5 mg/kg/time of ZKAB001 IV bi-weekly. DLT will be observed within 28 days after administration.
  Interventions: Drug: ZKAB001 5mg/kg
- ZKAB001 10mg/kg (Experimental): Three or six patients will be treated with the dose of 5 mg/kg/time of ZKAB001 IV bi-weekly. DLT will be observed within 28 days after administration.
  Interventions: Drug: ZKAB001 10mg/kg
- ZKAB001 15mg/kg (Experimental): Three or six patients will be treated with the dose of 5 mg/kg/time of ZKAB001 IV bi-weekly. DLT will be observed within 28 days after administration.
  Interventions: Drug: ZKAB001 15mg/kg

INTERVENTIONS:
Drug: ZKAB001 5mg/kg — 5mg/kg/times bi-week IV administration of ZKAB001
  Other Names: PD-L1 monoclonal antibody
  Arms: ZKAB001 5mg/kg
Drug: ZKAB001 10mg/kg — 10mg/kg/times bi-week IV administration of ZKAB001
  Other Names: PD-L1 monoclonal antibody
  Arms: ZKAB001 10mg/kg
Drug: ZKAB001 15mg/kg — 15mg/kg/times bi-week IV administration of ZKAB001
  Other Names: PD-L1 monoclonal antibody
  Arms: ZKAB001 15mg/kg

SUMMARY:
This is a Phase 1+2, open-label, dose-escalation, and multidose study, aiming to investigate the safety, tolerability and pharmacokinetics of ZKAB001 (a fully human monoclonal antibody targeting the Programmed Death - Ligand 1 (PD-L1) membrane receptor on T lymphocytes and other cells of the immune system) administered every 14 days in subjects with locally advanced and metastatic urothelial carcinoma.

DETAILED DESCRIPTION:
The study will consist of 4 periods: Screening (up to 28 days), Lead-in period (Day -28), Treatment (up to 24 cycles or 1 year, whichever occurs first）, and Follow-up (up to 1 year). There will be a lead-in period on Day -28 for each dose escalation cohort in which the single-dose pharmacokinetics(PK) of ZKAB001 will be characterized prior to initiation of continuous dosing in the first cycle of treatment. The lead-in period duration, PK time-points, doses and/or regimens used in subsequent cohorts may be modified based on the exposure (AUC) observed during the lead-in period (although the number of PK samples will not be increased). Treatment of continuous dosing is up to 24 cycles or 1 year, until as per investigator's opinion, subjects experience disease progression (evaluated by RECIST 1.1 and immune-related response criteria irRECIST), no clinical benefit, or intolerable toxicity. If investigators suspect subjects experience pseudoprogression or has evidence to prove "mixed response", subjects can continue to accept treatment as investigator decided.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily gives written informed consent to participate in the study.
2. Female and male patients aged between 18 and 75 (inclusive).
3. Subjects must have a histologically and/or cytologically confirmed diagnosis of urothelial carcinoma and the recurrence or metastasis is confirmed again after recurrence, and must have failed or are intolerable to standard therapies or for whom no standard therapies exist.
4. Must have measurable disease with at least 1 unidimensional measurable lesion (recorded as the maximum diameter) based on RECIST 1.1.
5. Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1, with estimated life expectancy of at least 3 months.
6. Adequate blood routine, hepatic and renal function:

1)neutrophil count (ANC) absolutely acuity≥1.5 x 109 / L; 2)platelet count≥80 x 109 / L ; 3)hemoglobin≥90 g/L; 4)serum albumin≥28 g/L; 5)bilirubin≤1.5 x ULN (upper limit of normal ); 6)ALT and AST≤1.5 x ULN, such as liver metastasis, ALT (alanine transaminase) and AST≤5 x ULN; 7)serum Cr≤1.25 x ULN or endogenous creatinine clearance≥50 ml/min (according Cockcroft Gault formula).

7.Female patients of reproductive age should take effective contraception during the study period and within 3 months after the study treatment period. The serum or urine human chorionic gonadotropin (HCG) examination must be negative within 7 days before the study was enrolled.

Exclusion Criteria:

1. Any active autoimmune disease or history of autoimmune disease (such as, but not limited to, interstitial pneumonia, uveitis, enteritis, hepatitis, arthritis, nephritis, pituitary inflammation, hyperthyroidism, hypothyroidism, etc.); Patients with vitiligo or asthma in childhood, and still need medical intervention in adult; Patients need bronchodilators for medical intervention of asthma.
2. Patients are using immunosuppressive agents, or systemic, or absorbable topical corticosteroid medications to achieve immunosuppressive purposes (doses >10mg/day prednisone or equivalent), which is ongoing 2 weeks before enrollment.
3. Have received any form of organ transplantation, including allogeneic stem cell transplantation.
4. Known allergy to macromolecular protein inhibitors or any of the components of ZKAB001.
5. Suffering from other malignant tumors other than this diseases in 5 years except skin basal cell and squamous cell carcinoma or cervical carcinoma in situ.
6. Central nervous system metastases with clinical symptoms (such as cerebral edema and brain metastases requiring corticosteroid intervention). Previous treatment with brain or meningeal metastasis, such as clinical stabilization (MRI) less than 2 months, or systemic corticosteroid (dose >10mg/day prednisone or equivalent) less than 2 weeks.
7. Patients with clinical symptoms or heart diseases that cannot be well controlled, such as heart failure above New York Heart Association (NYHA) 2 grade, unstable angina pectoris, myocardial infarction in 1 year, and clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention, left ventricular ejection fraction < 50% at rest as shown in the ultrasound cardiogram.
8. Patients who had received radiotherapy, chemotherapy, surgery or molecular targeted therapy before, were given less than 4 weeks or 5 half-life (longer time) after the treatment (if treated with nitrosourea or mitomycin previously, the time interval between the end of chemotherapy and study inclusion was less than 6 weeks); Adverse events caused by previous treatment did not recover to level 1 of CTCAE, except for hair loss.
9. Active infection, or unexplained fever> 38.5 degrees during screening period or before the first dose of ZKAB001 (subjects with fever from the tumor could be enrolled upon investigator's decision).
10. Human immunodeficiency virus (HIV) positive, syphilis spirochete positive, untreated active hepatitis.
11. The patient is participating in other clinical studies or is less than 1 month away from the end of the previous clinical study.
12. Patients may need to receive other systemic cancer treatment during study period.
13. Prior therapy with an anti-PD 1, anti-PD L1, or anti-CTLA-4 (Cytotoxic T Lymphocyte Antigen-4) antibody (or any other agents that target immunoregulatory receptor).
14. Recent history of prophylactic non-cancer vaccination (such as seasonal influenza vaccine and human papillomavirus (HPV) vaccine) within 28 days before screening.
15. History of mental drug abuse, alcohol abuse or drug abuse.
16. Pregnant or lactating women.
17. Any mental condition that prevents the understanding or provision of an informed consent.
18. It is determined by the investigator that the patient has other factors that may lead to the termination of the study, such as other serious diseases or serious laboratory test abnormalities or other factors that may affect the safety of the subjects, family or social factors that may affect the study data and sample collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-10-10 (Estimated); Primary Completion 2020-02-14 (Estimated); Study Completion 2023-06-23 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days after first dose
  Adverse events of level 3 or above related to the study drug occurring within 28 days after the first dose as assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Maximal tolerable dose(MTD) | 28 days after first dose
  DLT occurs in less than 1/6 subjects, this lower dose is defined as MTD.
The overall response rate(ORR) | through study completion, an average of 2 year
  The proportion of subjects who achieve the optimal objective response rate (PR or CR).
AUC(0-t) | 24 periods or 1 year
  Area under curve 0-t
AUC(INF) | 24 periods or 1 year
  Area under curve INF
Cmax | 24 periods or 1 year
  Peak concentration
Tmax | 24 periods or 1 year
  Peak time
T1/2 | 24 periods or 1 year
  Half life
Vss | 24 periods or 1 year
  Steady-state apparent volume of distribution based on plasma concentration
Total body clearance(CLT) | 24 periods or 1 year
  Total body clearance
Cmin | 24 periods or 1 year
  The trough value at steady state
The percentage of the receptors of PD-L1 in CD14+(cluster of differentiation 14+) monocytes and CD3+(cluster of differentiation 3+) T cells | through study completion, an average of 2 year
  To detected the percentage of the receptors of PD-L1 in CD14+ monocytes and CD3+ T cells.
The number of subjects presenting detectable anti drug antibodies (ADAs) | through study completion, an average of 2 year
  To evaluated the number of subjects presenting detectable anti drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Study Director — Beijing Tumor Hospital
Locations (1):
- Beijing Tumor Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No